CLINICAL TRIAL: NCT04220489
Title: Perioperative Ketamine in Opioid-Tolerant Patients Undergoing Lumbar Spine Surgery: A Randomized, Double-blind, Placebo-controlled Trial
Brief Title: Perioperative Ketamine in Opioid-Tolerant Patients Undergoing Lumbar Spine Surgery
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study stopped due to unexpected issues surrounding the 2020 COVID-19 pandemic
Sponsor: Jacques E. Chelly (Other)
Responsible Party: Sponsor-Investigator, Jacques E. Chelly, Professor of Anesthesiology and Perioperative Medicine and Orthopedic Surgery Director, Regional Anesthesiology Fellowship Program, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STUDY19020144
Record Dates: First submitted 2019-11-21; First posted 2020-01-07 (Actual); Results first posted 2024-01-30 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Opioid Dependence; Chronic Pain
Keywords: Ketamine; Lumbar Spine Surgery; Opioid Tolerant
MeSH Terms: conditions — Opioid-Related Disorders; Chronic Pain | interventions — Ketamine

STUDY DESIGN:
Intervention Model Description: Prospective, Randomized, Double-Blind, Placebo Controlled trial involving opiate-dependent patients undergoing lumbar spine surgery
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ketamine Group (Experimental): Participants will receive a 1 mg/kg dose of intravenous ketamine 15 minutes after induction of general anesthesia. Thereafter, a continuous infusion of 0.20 mg/kg/hr ketamine with a maximum dose of 20 mg/hr will be run to conclude at 48 hours after the end of the surgery (fascial closure).
  Interventions: Drug: Ketamine
- Placebo Group (Placebo Comparator): Participants will receive a 1 mg/kg dose of intravenous saline 15 minutes after induction of general anesthesia. Thereafter, a continuous infusion of 0.20 mg/kg/hr saline with a maximum dose of 20 mg/hr will be run to conclude at 48 hours after the end of the surgery (fascial closure).
  Interventions: Drug: Placebo Comparator

INTERVENTIONS:
Drug: Ketamine — Intraoperative ketamine and post operative 48 hour ketamine infusion with a standardized general anesthesia protocol.
  Other Names: Ketalar
  Arms: Ketamine Group
Drug: Placebo Comparator — Participants will receive a 1 mg/kg dose of intravenous saline 15 minutes after induction of general anesthesia. Thereafter, a continuous infusion of 0.20 mg/kg/hr saline with a maximum dose of 20 mg/hr will be run to conclude at 48 hours after the end of the surgery (fascial closure)
  Other Names: Placebo Group
  Arms: Placebo Group

SUMMARY:
The goal of this study is to determine whether comprehensive perioperative administration of the N-methyl-D-aspartate (NMDA) receptor antagonist ketamine can increase postoperative pain tolerance and reduce opiate consumption in chronic back pain patients undergoing spinal laminectomy/fusion when compared to placebo

Opioid dependence will be defined as daily opioid use (2 or more doses per day) for a period of two-months or longer. Intraoperatively, patients will receive a 1 mg/kg dose of intravenous ketamine or saline with 15 minutes after induction of general anesthesia. Thereafter, a continuous infusion of 0.20 mg/kg/hr ketamine with a maximum dose of 20 mg/hr or saline will be run to conclude at 24 hours after the end of the surgery (fascial closure). The primary outcome measure will be hydromorphone PCA usage during the first 72 hours postoperatively. Secondary outcome measures will be VAS pain scores at rest and with movement in PACU, 24 hr, 48 hr, 72 hr, 2 week (post-op visit), 6 week follow-up visit, as well as, McGill Pain Questionnaire, Pain Catastrophizing Scale, and emotional distress surveys assessing depression and anxiety at preop/screening, postop and 6 week follow-up (PROMIS Emotional Distress-Anxiety Short Form, PROMIS Emotional Distress-Depression Short Form), as well as a Neuro-QOL Short Form v1.1 - Satisfaction with Social Roles and Activities .

DETAILED DESCRIPTION:
Patients will be recruited from the University of Pittsburgh Medical Center (UPMC) Neurosurgery Clinic and Operating Room Schedule. The primary surgeon will identify patients who would be eligible for inclusion, ask them if they would be interested in participating, and if so, the enrollment and consent process would be initiated. The participating neurosurgeons include Dr. Okonkwo and Dr. Hamilton, who have agreed to allow us access to their patients. Informed consent will be performed by the surgeon or the PI. Enrollment will be performed by the study coordinator and/or trained representative from the Acute Interventional Perioperative Pain Service (AIPPS). Enrollment will include review of eligibility, and detailed explanation of the study.

Screening Visit:

After patients are enrolled into the study at the preoperative neurosurgery clinic, a number of forms will be filled out by the participants: McGill Pain questionaire-Short form, pain medication review form, and the Pain Catastrophizing Scale (PCS) (Sullivan, 1995). PROMIS Emotional Distress-Anxiety Short Form and PROMIS Emotional Distress-Depression Short Form, Brief Psychiatric Rating Scale and Neuro-QoL Short Form v1.1 - Satisfaction with Social Roles and Activities will also be completed.

Pre-Operative Visit:

The participant will be asked to come into the Aiken Medical Building, Suite 407 on a date after the clinic visit but before their day of surgery for a Pre-Operative Visit. Investigators will work with the participant to determine their opioid dose regimen, and the participant will be asked to come into the Aiken Medical Building thirty minutes before their opioid dose is due and will be asked to bring with them their upcoming dose of pain medication. Prior to taking their pain medication, the participant will then be administered a cold-pressor pain sensitivity test. Heart rate and blood pressure will be recorded before and after the cold-pressor test. Once the cold pressor test is completed, the McGill Pain Questionnaire will be administered. After this questionnaire is complete, the participant will take the dose of opioid medication they have brought from home and are scheduled to receive and will wait in the clinic for 30 minutes for the pain medication to take effect. Once the 30 minutes is complete, the cold-pressor test will be repeated, heart rate and blood pressure collected before and after, and McGill Pain Questionnaire will be administered again.

Surgical Visit:

At the day of surgery, participants will be seen by team members of the Acute Interventional Perioperative Pain Service preoperatively. Patients will be randomized into the Ketamine Group or the Placebo Group.

A standardized general anesthesia protocol will be used by the hands-on provider. All drugs used intraoperatively, including total hydromorphone dose, will be collected from the electronic chart.

The amount of narcotics and non-narcotic analgesics administered in the operative and postoperative period will be collected from the electronic chart from day of surgery until discharge. Visual Analogue Scale (VAS) pain scores will be collected.

Post-Op Visit:

Patients will follow-up at Neurosurgery clinic at 10-14 days postoperatively. At this time daily opioid usage will be assessed and converted to morphine equivalents/24 hr. At this visit: pain medication review form, and the Pain Catastrophizing Scale (PCS) (Sullivan, 1995). PROMIS Emotional Distress-Anxiety Short Form and PROMIS Emotional Distress-Depression Short Form, Brief Psychiatric Rating Scale and Neuro-QoL Short Form v1.1 - Satisfaction with Social Roles and Activities will also be completed by the participant.

6-Week Follow-Up Visit:

The participant will be asked to come to the Aiken Medical Building, Suite 407 approximately 6 weeks after their surgery. Investigators will work with the participant to determine their post-operative opioid dose regimen. Prior to taking their pain medication, the participant will then be administered a cold-pressor pain sensitivity test, in a manner identical to that use during the pre-operative assessment.In addition to the McGill Pain Questionnaire-Short form, a pain medication review form, the Pain Catastrophizing Scale (PCS) (Sullivan, 1995), the PROMIS Emotional Distress-Anxiety Short Form, the PROMIS Emotional Distress-Depression Short Form, Brief Psychiatric Rating Scale and Neuro-QoL Short Form v1.1 - Satisfaction with Social Roles and Activities will also be completed.

ELIGIBILITY:
Inclusion Criteria

* Patients undergoing lumbar, thoracic or cervical spine surgery of at least one level, and no more than 6 levels.
* Patients with chronic back pain (>3 months)
* Anaesthetic risk assessment (ASA) 1-3
* Opiate-dependent with daily opiate use for at least 2 months and regimented daily narcotic dose twice a day/bis in die (BID) or greater or use of a regimented opioid pump

Exclusion Criteria

* Intolerance or known allergy to ketamine
* History of increased intraocular pressure (> 22mmHg)
* Uncontrolled hypertension (systolic blood pressure greater than or equal to 180, diastolic blood pressure greater than equal to 100)
* Increased intracranial pressure
* History of psychosis
* Pregnancy
* Patients with significant liver disease {signs and symptoms of liver injury, such as discolored skin and eyes that appear yellowish, abdominal pain and swelling, Itchy skin that doesn't seem to go away, dark urine color, pale stool color, bloody or tar-colored stool, chronic fatigue, nausea, loss of appetite, with or without elevated Liver Function Tests (LFTs): aspartate aminotransferase (AST) > 120 IU/ml, alkaline phosphatase (AP) >130 IU/ml, and alanine aminotransferase (ALT) >40 IU/ml}
* Patients with exposure to Cytochrome P450, family 3, subfamily A (CYP3A) and / or Cytochrome P450 Family 2 Subfamily B Member 6 (CYP2B6) inhibitors, including the herbs and the over-the-counter compounds (list of drugs can be found at http://www.fda.gov/drugs/developmentapprovalprocess/developmentresources/druginteractionslabeling/ucm093664.htm)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2019-12-17 (Actual); Primary Completion 2022-11-19 (Actual); Study Completion 2022-11-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jacques E Chelly, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- Jacques E Chelly, MD, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
There is no current plan to share individual participant data. In the future, the investigators may decide to share data with other investigators both within and outside of this institution. If that were to occur, we would de-identify all of the information prior to sharing any data in this way.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ketamine Group | Placebo Group
Started | 1 | 0
Completed | 1 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Only one subject was enrolled into this trial and they were in the ketamine group
Groups:
- Total: Total of all reporting groups
Arm/Group | Ketamine Group | Placebo Group | Total
Number analyzed (Participants) | 1 | 0 | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 0 | 1
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 44 (0.0) |  | 44 (0.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 |  | 0
  Male | 1 |  | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  | 0
  Asian | 0 |  | 0
  Native Hawaiian or Other Pacific Islander | 0 |  | 0
  Black or African American | 0 |  | 0
  White | 1 |  | 1
  More than one race | 0 |  | 0
  Unknown or Not Reported | 0 |  | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1 |  | 1

OUTCOME MEASURES:

1. Primary Outcome: Post-surgical Hydromorphone Patient Care Assistance (PCA) Opioid Utilization
Description: Hydromorphone Patient Care Assistant (PCA) usage during the first 72 hours postoperatively will be recorded. Hydromorphone opioid usage will be assessed and converted to morphine equivalents/24 hour. The higher the values, the worse the outcomes.
Time Frame: 72 hours postoperatively
Population: Only one subject was enrolled in this study and they were assigned to the ketamine group, therefore, no subjects are analyzed in the placebo group
Measure: Mean (Standard Deviation); unit: mg morphine equivalents per 24 hours
Arm/Group | Ketamine Group | Placebo Group
Number analyzed (Participants) | 1 | 0
mg morphine equivalents per 24 hours | 40 (0) |

2. Primary Outcome: Post-surgical Pain Rating Using the Visual Analog Scale (VAS)
Description: Post-surgical pain ratings will be measured by the assessment of participant's answers to the Visual Analog Scale (VAS). This measurement is a visual scale from 0-10, 0 being no pain, 5 being moderate pain and 10 being the worst imaginable pain. The lowest possible score is 0 and the highest possible score is 10. The participant will be asked to score pain at its best and worst over the period since they were last asked. Higher scores present a worse outcome. Pain will be monitored every four hours from the time the participant enters the PACU until discharge from the hospital, except during the night when the participant is asleep. The value reported consists of the average of all pain scores collected.
Time Frame: 72 hours post-operatively
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ketamine Group | Placebo Group
Number analyzed (Participants) | 1 | 0
units on a scale | 5 (0) |

3. Primary Outcome: Post-surgical Opioid Utilization Using Electronic Medication Review
Description: Post-surgical opioid utilization will be measured by reviewing participant's electronic medical records and recording opioid usage. Daily opioid usage will be assessed and converted to morphine equivalents/24 hr. The higher the values, the worse the outcomes.
Time Frame: 72 hours post-operatively
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg morphine equivalents per 24 hours
Arm/Group | Ketamine Group | Placebo Group
Number analyzed (Participants) | 1 | 0
mg morphine equivalents per 24 hours | 40 (0) |

4. Primary Outcome: Post-surgical Opioid Utilization Using Electronic Medication Review
Description: as for outcome 3
Time Frame: 6-week follow-up visit
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Ketamine Group | Placebo Group
Number analyzed (Participants) | 1 | 0
mg | 4 (0) |

5. Primary Outcome: Pre-surgical Opioid Utilization Using the Pain Medication Review Form
Description: Pre-surgical opioid utilization will be measured by the Pain Medication Review Form where patients will record all of the medications they are currently taking.
Time Frame: Screening visit
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: count of prescription medications
Arm/Group | Ketamine Group | Placebo Group
Number analyzed (Participants) | 1 | 0
count of prescription medications | 4 (0) |

6. Primary Outcome: Pre-surgical Pain Rating Using the Visual Analog Scale (VAS)
Description: Post-surgical pain ratings will be measured by the assessment of participant's answers to the Visual Analog Scale (VAS). This measurement is a visual scale from 0-10, 0 being no pain, 5 being moderate pain and 10 being the worst imaginable pain. The lowest possible score is 0 and the highest possible score is 10. Higher scores present a worse outcome.
Time Frame: Screening visit
Population: Data was not collected
Arm/Group | Ketamine Group | Placebo Group
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Pre-surgical Emotional Distress Related to Depression
Description: Pre-surgical emotional distress related to depression will be measured by assessment of participant's answers to the PROMIS Emotional Distress-Depression Short Form questionnaire. There are 8 questions about how the participant may have felt in the past 7 days. The scale is from 1, never have felt this way in the past 7 days, to 5, always have felt this way in the past 7 days. The questionnaire scores can be from a range of 8 being the least severe score and 40 being the most severe score. Higher scores present a worse outcome.
Time Frame: Screening visit
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ketamine Group | Placebo Group
Number analyzed (Participants) | 1 | 0
score on a scale | 27 (0) |

8. Secondary Outcome: Post-surgical Emotional Distress Related to Depression
Description: Post-surgical emotional distress related to depression will be measured by assessment of participant's answers to the PROMIS Emotional Distress-Depression Short Form questionnaire. There are 8 questions about how the participant may have felt in the past 7 days. The scale is from 1, never have felt this way in the past 7 days, to 5, always have felt this way in the past 7 days. The questionnaire scores can be from a range of 8 being the least severe score and 40 being the most severe score. Higher scores present a worse outcome. The value reported consists of the average of all questionnaire scores collected between POD 10 and POD 14.
Time Frame: Day 10-14 Post-Operative Visit
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ketamine Group | Placebo Group
Number analyzed (Participants) | 1 | 0
score on a scale | 14 (0) |

9. Secondary Outcome: Post-surgical Emotional Distress Related to Depression
Description: Post-surgical emotional distress related to depression will be measured by assessment of participant's answers to the PROMIS Emotional Distress-Depression Short Form questionnaire. There are 8 questions about how the participant may have felt in the past 7 days. The scale is from 1, never have felt this way in the past 7 days, to 5, always have felt this way in the past 7 days. The questionnaire scores can be from a range of 8 being the least severe score and 40 being the most severe score. Higher scores present a worse outcome.
Time Frame: 6-week follow-up visit
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ketamine Group | Placebo Group
Number analyzed (Participants) | 1 | 0
score on a scale | 19 (0) |

10. Secondary Outcome: Pre-surgical Emotional Distress Related to Anxiety
Description: Pre-surgical emotional distress related to anxiety will be measured by assessment of participant's answers to the PROMIS Emotional Distress-Anxiety Short Form questionnaire. There are 7 questions about how the participant may have felt in the past 7 days. The scale is from 1, never have felt this way in the past 7 days, to 5, always have felt this way in the past 7 days. The questionnaire scores can be from a range of 7 being the least severe score and 35 being the most severe score. Higher scores present a worse outcome.
Time Frame: Screening visit
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ketamine Group | Placebo Group
Number analyzed (Participants) | 1 | 0
score on a scale | 23 (0) |

11. Secondary Outcome: Post-surgical Emotional Distress Related to Anxiety
Description: Post-surgical emotional distress related to anxiety will be measured by assessment of participant's answers to the PROMIS Emotional Distress-Anxiety Short Form questionnaire. There are 7 questions about how the participant may have felt in the past 7 days. The scale is from 1, never have felt this way in the past 7 days, to 5, always have felt this way in the past 7 days. The questionnaire scores can be from a range of 7 being the least severe score and 35 being the most severe score. Higher scores present a worse outcome. The value reported consists of the average of all questionnaire scores collected between POD 10 and POD 14.
Time Frame: Day 10-14 Post-Operative Visit
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ketamine Group | Placebo Group
Number analyzed (Participants) | 1 | 0
score on a scale | 16 (0) |

12. Secondary Outcome: Post-surgical Emotional Distress Related to Anxiety
Description: Post-surgical emotional distress related to anxiety will be measured by assessment of participant's answers to the PROMIS Emotional Distress-Anxiety Short Form questionnaire. There are 7 questions about how the participant may have felt in the past 7 days. The scale is from 1, never have felt this way in the past 7 days, to 5, always have felt this way in the past 7 days. The questionnaire scores can be from a range of 7 being the least severe score and 35 being the most severe score. Higher scores present a worse outcome.
Time Frame: 6-week follow-up visit
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ketamine Group | Placebo Group
Number analyzed (Participants) | 1 | 0
score on a scale | 19 (0) |

13. Secondary Outcome: Pre-surgical Satisfaction With Social Roles and Activities
Description: Pre-surgical satisfaction with social roles and activities will be measured by assessment of participant's answers to the Neuro-QoL Short Form v1.1 - Satisfaction with Social Roles and Activities questionnaire. There are 8 questions about how the participant may have felt in the past 7 days. The scale is from 1, never have felt this way in the past 7 days, to 5, always have felt this way in the past 7 days. The questionnaire scores can be from a range of 8 being the least satisfaction score and 40 being the most satisfaction score. Higher scores present a better outcome.
Time Frame: Screening visit
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ketamine Group | Placebo Group
Number analyzed (Participants) | 1 | 0
score on a scale | 19 (0) |

14. Secondary Outcome: Post-surgical Satisfaction With Social Roles and Activities
Description: Post-surgical satisfaction with social roles and activities will be measured by assessment of participant's answers to the Neuro-QoL Short Form v1.1 - Satisfaction with Social Roles and Activities questionnaire. There are 8 questions about how the participant may have felt in the past 7 days. The scale is from 1, never have felt this way in the past 7 days, to 5, always have felt this way in the past 7 days. The questionnaire scores can be from a range of 8 being the least satisfaction score and 40 being the most satisfaction score. Higher scores present a better outcome. The value reported consists of the average of all questionnaire scores collected between POD 10 and POD 14.
Time Frame: Day 10-14 Post-Operative Visit
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ketamine Group | Placebo Group
Number analyzed (Participants) | 1 | 0
score on a scale | 21 (0) |

15. Secondary Outcome: Post-surgical Satisfaction With Social Roles and Activities
Description: Post-surgical satisfaction with social roles and activities will be measured by assessment of participant's answers to the Neuro-QoL Short Form v1.1 - Satisfaction with Social Roles and Activities questionnaire. There are 8 questions about how the participant may have felt in the past 7 days. The scale is from 1, never have felt this way in the past 7 days, to 5, always have felt this way in the past 7 days. The questionnaire scores can be from a range of 8 being the least satisfaction score and 40 being the most satisfaction score. Higher scores present a better outcome.
Time Frame: 6-week follow-up visit
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ketamine Group | Placebo Group
Number analyzed (Participants) | 1 | 0
score on a scale | 20 (0) |

16. Secondary Outcome: Pre-surgical Pain Rating Using the Pain Catastrophizing Scale
Description: Pre-surgical pain ratings will be measured by the assessment of participant's answers to the Pain Catastrophizing Scale questionnaire. There are 14 statements related to pain that participants will record experiencing on a scale of 0 being experienced not at all to 4 being experienced all of the time. The lowest possible score is 0 and the highest possible score is 56. Higher scores present a worse outcome.
Time Frame: Screening visit
Population: Data not collected
Arm/Group | Ketamine Group | Placebo Group
Number analyzed (Participants) | 0 | 0

17. Secondary Outcome: Post-surgical Pain Rating Using the Pain Catastrophizing Scale
Description: Post-surgical pain ratings will be measured by the assessment of participant's answers to the Pain Catastrophizing Scale questionnaire. There are 14 statements related to pain that participants will record experiencing on a scale of 0 being experienced not at all to 4 being experienced all of the time. The lowest possible score is 0 and the highest possible score is 56. Higher scores present a worse outcome
Time Frame: Day 10-14 Post-Operative Visit
Population: Data not collected
Arm/Group | Ketamine Group | Placebo Group
Number analyzed (Participants) | 0 | 0

18. Secondary Outcome: Post-surgical Pain Rating Using the Pain Catastrophizing Scale
Description: as for outcome 17
Time Frame: 6-week follow-up visit
Population: Data not collected
Arm/Group | Ketamine Group | Placebo Group
Number analyzed (Participants) | 0 | 0

19. Secondary Outcome: Pre-surgical Opioid Analgesic Efficacy Using the Cold-Pressor Pain Sensitivity Test
Description: Pre-surgical opioid analgesic efficacy will be measured by the results of the Cold-Pressor Pain Sensitivity Test, where the participant will submerge their hand in ice water for up to four minutes at thirty minutes before and thirty minutes after the participant's opioid pain medication is taken. Pain tolerance is defined as the time in seconds that it takes for the participant to withdraw their hand from the ice water. Pain threshold, tolerance and cut-off will be recorded using a stopwatch. The McGill Pain Questionnaire short form will be completed after each test. Opioid-analgesic efficacy will be estimated by the change in pain threshold and tolerance observed after the opioid was consumed relative to initial assessment of pain threshold and tolerance. The higher the tolerance after opioid consumption, the better the outcomes.
Time Frame: Screening visit
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Ketamine Group | Placebo Group
Number analyzed (Participants) | 1 | 0
seconds | 19.49 (0.98) |

20. Secondary Outcome: Post-surgical Opioid Analgesic Efficacy Using the Cold-Pressor Pain Sensitivity Test
Description: Post-surgical opioid analgesic efficacy will be measured by the results of the Cold-Pressor Pain Sensitivity Test, where the participant will submerge their hand in ice water for up to four minutes at thirty minutes before and thirty minutes after the participant's opioid pain medication is taken. Pain tolerance is defined as the time in seconds that it takes for the participant to withdraw their hand from the ice water. Pain threshold, tolerance and cut-off will be recorded using a stop watch. The McGill Pain Questionnaire short form will be completed after each test. Opioid-analgesic efficacy will be estimated by the change in pain threshold and tolerance observed after the opioid was consumed relative to initial assessment of pain threshold and tolerance. The higher the threshold and tolerance after opioid consumption, the better the outcomes.
Time Frame: 6-week follow-up visit
Population: Data not collected
Arm/Group | Ketamine Group | Placebo Group
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of signed consent to 6-weeks
Description: The placebo group has 0 participants at risk, since no participants were enrolled into this group
Arm/Group | Ketamine Group | Placebo Group
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/0
Other Adverse Events (participants affected / at risk) | 0/1 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (3):
  • Study Protocol (2019-09-03): https://cdn.clinicaltrials.gov/large-docs/89/NCT04220489/Prot_000.pdf
  • Statistical Analysis Plan (2019-09-03): https://cdn.clinicaltrials.gov/large-docs/89/NCT04220489/SAP_001.pdf
  • Informed Consent Form (2022-01-04): https://cdn.clinicaltrials.gov/large-docs/89/NCT04220489/ICF_002.pdf